CLINICAL TRIAL: NCT00465608
Title: Reduction of the Traumatic Memory by Reconsolidation Blockade: A Pilot Study
Brief Title: Propranolol in Post Traumatic Stress Disorder
Acronym: Reductrauma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: M.E. Llau, UHToulouse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0604603
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: adults; PTSD; trauma; AZF; propranolol; reconsolidation; Post traumatic stress disorder; chronic form; PTSD (Post-Traumatic Stress Disorder)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Combat Disorders | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): propranolol
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — propranolol by mouth (per os)
  Other Names: betablocker

SUMMARY:
Problem and Objectives: There is currently no pharmacological treatment for curing post traumatic stress disorder (PTSD). The investigators will test whether propranolol when given immediately after trauma evocation is able to decrease the strength of the traumatic memory, and by extension, the severity of PTSD symptoms associated with that memory.

Hypotheses:

1. The subjects will show a significant pre/post decrease in PTSD symptoms.
2. Those gains will be maintained at follow-up.

Study Design: Open pharmacological trial.

Method: On the first visit (V1), the subjects will describe their traumatic experience in writing and will receive the propranolol. A script describing this experience will be constructed to be used in the subsequent encounters to elicit the trauma memory. A week later (V2), before receiving the propranolol, subjects will be asked to read aloud their trauma script while imagining it as vividly as possible for 10 minutes. This weekly treatment will be repeated 6 times (from V1 to V6). A total of 6 doses of propranolol will be given. A self-report measure will be used to monitor improvement in PTSD symptomatology on the following visits: V1, V4, V6, V7 and V8 (3 month follow-up).

Statistical Analyses: A repeated measure ANOVA (pre-test, post-test, and 3-month follow-up) using the PTSD symptom score will be conducted.. Three t-tests will be performed to examine simple effects. The alpha level will be set at p = .05 (two-tailed). Fisher's exact test will be used to examine whether Ss still meet the diagnostic criteria for PTSD at the end of the study.

Clinical Implications: If this treatment is effective, a randomized controlled trial will be launched. This treatment has the potential to become the first pharmacological treatment designed to cure PTSD.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Suffer from AZF-related PTSD (PCL score more than 44)
* Sign consent form
* Subjects must have health coverage.

Exclusion Criteria:

* Not diagnosed with current, chronic AZF-related PTSD
* Age < 18 or > 65
* Systolic blood pressure < 100 mm Hg
* Medical condition that contraindicates the administration of propranolol, e.g., history of congestive heart failure, heart block, insulin-requiring diabetes, chronic bronchitis, emphysema, or asthma. With regard to asthma, because many persons who say they have had an asthma attack, especially as a child, may only have had hay fever, another allergy, or another non-asthmatic episode, a blanket exclusion criterion may be overly restrictive. Therefore, asthma attacks will only be exclusionary if they:

  * occurred within the past ten years,
  * occurred at any time in life if induced by a β-blocker, or
  * are currently being treated, regardless of the date of last occurrence.

Cardiological consultation will be obtained as necessary.

* Previous adverse reaction to, or non-compliance with, a β-blocker
* Current use of medication that may involve potentially dangerous interactions with propranolol, including, other β-blockers, antiarrhythmics, calcium channel blockers, and potent P450 2D6 inhibitors, e.g., fluoxetine, paroxetine, miconazole, sulconazole, metoclopramide, quinidine, ticlopidine, and ritonavir.
* Contraindicating psychiatric condition, including lifetime or current psychotic, bipolar, melancholic, or substance dependence or abuse disorder; suicidality.
* Initiation of, or change in, psychotropic medication within the previous two months. For subjects receiving stable doses of pharmacotherapy, they and their providers will be asked not to change the regimen except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the subject or terminating participation.
* Current participation in any psychotherapy (other than strictly supportive). Subjects will be asked not to initiate psychotherapy during the course of the proposed study except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis with regard to retaining the subject or terminating participation.
* Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation
* Does not understand French

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist score | 3 months

SECONDARY OUTCOMES:
SCID diagnosis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIRMES, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Psychiatric Department, Toulouse, France

REFERENCES:
- [Background] Pitman RK, Sanders KM, Zusman RM, Healy AR, Cheema F, Lasko NB, Cahill L, Orr SP. Pilot study of secondary prevention of posttraumatic stress disorder with propranolol. Biol Psychiatry. 2002 Jan 15;51(2):189-92. doi: 10.1016/s0006-3223(01)01279-3. PMID 11822998
- [Background] Vaiva G, Ducrocq F, Jezequel K, Averland B, Lestavel P, Brunet A, Marmar CR. Immediate treatment with propranolol decreases posttraumatic stress disorder two months after trauma. Biol Psychiatry. 2003 Nov 1;54(9):947-9. doi: 10.1016/s0006-3223(03)00412-8. PMID 14573324